CLINICAL TRIAL: NCT01169337
Title: Randomized Phase III Trial of Lenalidomide Versus Observation Alone in Patients With Asymptomatic High-Risk Smoldering Multiple Myeloma
Brief Title: Lenalidomide or Observation in Treating Patients With Asymptomatic High-Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02057; NCI-2011-02057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E3A06; CDR0000682012; E3A06 (Other: ECOG-ACRIN Cancer Research Group); E3A06 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Light Chain Deposition Disease; Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Watchful Waiting; Observation; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (lenalidomide) (Experimental): Patients receive lenalidomide PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm B (observation) (Active Comparator): Patients undergo observation until progression to symptomatic myeloma.
  Interventions: Other: Clinical Observation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm B (observation)
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm A (lenalidomide)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II/III trial studies how well lenalidomide works and compares it to observation in treating patients with asymptomatic high-risk asymptomatic (smoldering) multiple myeloma. Biological therapies such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Sometimes the cancer may not need treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether lenalidomide is effective in treating patients with high-risk smoldering multiple myeloma than observation alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the risk of grade 3 adverse events that effect vital organ function (such as cardiac, hepatic or thromboembolic) or any grade 4 or higher non-hematologic adverse events among patients receiving lenalidomide as treatment for high-risk asymptomatic, smoldering multiple myeloma. (Phase II) II. To compare progression free survival where failure is defined as death or the development of symptomatic myeloma indicating treatment between patients receiving lenalidomide versus observation alone in high-risk asymptomatic, smoldering multiple myeloma. (Phase III)

SECONDARY OBJECTIVES:

I. To assess the response to therapy of patients treated with lenalidomide as treatment for asymptomatic, smoldering multiple myeloma. (Phase II) II. To determine and compare the response rate, time to progression, 1-year progression-free survival probability, and overall survival between patients randomized to receive lenalidomide or observation in the setting of asymptomatic myeloma. (Phase III) III. To estimate the incidence of adverse events in patients receiving lenalidomide therapy for early-stage multiple myeloma. (Phase III)

CORRELATIVE OBJECTIVES:

I. To describe the cohort in terms of gene expression profiling (GEP) and cytogenetic risk classification and evaluate baseline immune and magnetic resonance imaging (MRI) parameters. (Phase II) II. To evaluate the impact of therapy within GEP-defined risk groups and GEP as a prognostic marker. (Phase III) III. To study the effects of lenalidomide on laboratory markers of immune function. (Phase III) IV. To study the prognostic value of MRI-detected asymptomatic bone disease on clinical outcome. (Phase III) V. To evaluate the prognostic effect of baseline high-risk cytogenetic abnormalities on clinical outcome. (Phase III)

QUALITY OF LIFE ASSESSMENT OBJECTIVES:

I. To compare quality of life (QOL) change between treatment and observation arms based on the functional (FWB) and physical (PWB) well-being components of the Functional Assessment of Cancer Therapy (FACT)-General (G) patient-reported outcome (PRO) measure from registration (prior to initiation of treatment) up to cycle 24.

II. To examine the impact of differential treatment response (PFS), if observed, on QOL based on the FACT FWB+PWB up to cycle 48.

III. To obtain prospective data on myeloma specific QOL attributes, utilizing and evaluating the Multiple Myeloma Subscale (MMS).

OUTLINE:

PHASE II: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE III: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive lenalidomide PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo observation until progression to symptomatic myeloma.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with asymptomatic high-risk smoldering multiple myeloma (SMM) within the past 60 months, as confirmed by both of the following:

  * Bone marrow plasmacytosis with >= 10% plasma cells or sheets of plasma cells at any time before initiating study treatment, including a marrow which must be obtained by bone marrow aspiration and/or biopsy within 4 weeks prior to randomization
  * Abnormal serum free light chain ratio (< 0.26 or > 1.65) by serum free light chain (FLC) assay; FLC assay must be performed within 28 days of randomization
* Patients must have measurable levels of monoclonal protein (M-protein): >= 1g/dL on serum protein electrophoresis or >= 200 mg of monoclonal protein on a 24 hour urine protein electrophoresis which must be obtained within 4 weeks prior to randomization
* Patients must have no lytic lesions on skeletal surveys and no hypercalcemia (i.e., >= 11 mg/dL)
* Hemoglobin >= 11 g/dL within four weeks prior to randomization
* Platelet count >= 100,000/mm^3 within four weeks prior to randomization
* Absolute neutrophil count (ANC) >= 1,500/mm^3 within four weeks prior to randomization
* Calculated creatinine clearance >= 30 mL/min within four weeks prior to randomization
* Bilirubin =< 1.5 mg/dL within four weeks prior to randomization
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGPT) (aspartate aminotransferase [AST]) =< 2.5 times upper limit of normal within four weeks prior to randomization
* No prior or concurrent systemic or radiation therapy for the treatment of myeloma
* Concurrent use of bisphosphonates is not permitted; however, prior bisphosphonates or once-a-year intravenous bisphosphonate given for the treatment of osteoporosis is permitted
* Prior or concurrent use of erythropoietin is disallowed
* Prior glucocorticosteroid therapy for the treatment of multiple myeloma is not permitted
* Prior systemic glucocorticosteroid use for the treatment of non-malignant disorders is permitted; concurrent use after registration on the study should be restricted to the equivalent of prednisone 10 mg per day
* Prior or concurrent topical or localized glucocorticosteroid therapy to treat non-malignant comorbid disorders is permitted
* Patients must not have active, uncontrolled seizure disorder; patients must have had no seizures in the last 6 months
* Patients must not have uncontrolled intercurrent illness including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation that would limit compliance with the study, or a prior history of Stevens Johnson syndrome
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Patients must not have baseline bone lesions or plasmacytomas
* Patients with monoclonal gammopathy of undetermined significance are not eligible
* Patients must not have grade 2 or higher peripheral neuropathy
* Patients must not have active, uncontrolled infection
* Patients may have a history of current or previous deep vein thrombosis or pulmonary embolism but are required to take some form of anti-coagulation as prophylaxis if they are not currently on full-dose anticoagulation
* Patients should not have New York Heart Association classification III or IV heart failure
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for the time period considered appropriate for cure of the specific cancer; for most diseases this time frame is 5 years
* Patients should not be felt to have an immediate need for chemotherapy
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting cycle 1 of lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Human immunodeficiency virus (HIV) infection is not excluded; HIV+ patients must meet the following criteria:

  * Cluster of differentiation (CD)4 cell count >= 350/mm^3
  * No history of acquired immune deficiency syndrome (AIDS)-related illness
  * Not currently prescribed zidovudine or stavudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Lonial, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (607):
- United States (603):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Saint Jude Medical Center, Fullerton, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - York Hospital, York Village, Maine
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Garnet Health Medical Center, Middletown, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Rutland Regional Medical Center, Rutland, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Ireland (3):
  - Mater Misericordiae University Hospital, Dublin, Co Dublin
  - Mater Private Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
- Fundacion De Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Lonial S, Jacobus S, Fonseca R, Weiss M, Kumar S, Orlowski RZ, Kaufman JL, Yacoub AM, Buadi FK, O'Brien T, Matous JV, Anderson DM, Emmons RV, Mahindra A, Wagner LI, Dhodapkar MV, Rajkumar SV. Randomized Trial of Lenalidomide Versus Observation in Smoldering Multiple Myeloma. J Clin Oncol. 2020 Apr 10;38(11):1126-1137. doi: 10.1200/JCO.19.01740. Epub 2019 Oct 25. PMID 31652094
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2011 and January 2013, 44 patients were enrolled in the phase II safety run in portion of the study and were treated with lenalidomide as a single agent. Between February 2013 and July 2017, 182 patients were randomly assigned between the two treatment arms in the phase III portion of the study.
Groups:
- Arm A (Lenalidomide; Phase II); Arm A (Lenalidomide; Phase III): Patients receive lenalidomide PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Observation; Phase III): Patients undergo observation until progression to symptomatic myeloma.
Period: Overall Study
Arm/Group | Arm A (Lenalidomide; Phase II) | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Started | 44 | 90 | 92
Received Treatment/Observation | 44 | 88 | 86
Completed | 0 | 0 | 86
Not Completed | 44 | 90 | 6
Not completed — Lack of Efficacy | 5 | 7 | 0
Not completed — Adverse Event | 12 | 18 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 11 | 6
Not completed — Noncompliance | 2 | 0 | 0
Not completed — Other complicating disease | 1 | 1 | 0
Not completed — Physician Decision | 1 | 5 | 0
Not completed — Alternative therapy | 0 | 2 | 0
Not completed — Changed hospital | 0 | 1 | 0
Not completed — Never started treatment | 0 | 2 | 0
Not completed — Reason not reported | 1 | 0 | 0
Not completed — Continuing lenalidomide | 9 | 43 | 0

BASELINE CHARACTERISTICS:
Population: All registered patients in phase II portion and randomized patients in phase III portion
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Lenalidomide; Phase II) | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III) | Total
Number analyzed (Participants) | 44 | 90 | 92 | 226
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 83] | 63 [31 to 82] | 64 [33 to 96] | 64 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 48 | 46 | 118
  Male | 20 | 42 | 46 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 6
  Not Hispanic or Latino | 43 | 81 | 81 | 205
  Unknown or Not Reported | 1 | 7 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 12 | 19 | 37
  White | 37 | 72 | 68 | 177
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Grade 3 Adverse Events That Effect Vital Organ Function or Any Grade 4 or Higher Non-hematologic Adverse Events (Phase II Primary Endpoint)
Description: Proportion of patients with grade 3 adverse events that effect vital organ function (such as cardiac, hepatic or thromboembolic) or any grade 4 or higher non-hematologic adverse events
Time Frame: Assessed every 4 weeks while on treatment up to 24 weeks
Population: The first 36 patients in the phase II part as planned in the study design
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase II)
Number analyzed (Participants) | 36
proportion of participants | 0.056 [0.010 to 0.165]

2. Primary Outcome: 2-year Progression-free Survival (PFS) Rate (Phase III Primary Endpoint)
Description: PFS is defined as time from randomization to progression or death, whichever occurs first. Patients are considered to have progression if both of the following criteria are met. Kaplan-Meier method was used to estimate 2-year PFS rate.
  1. Any of the following:
     * Increase in serum M-protein to ≥ 25% above the lowest response level with an absolute increase of at least 0.5g/dl to qualify as "progression"
     * Increase in urine M-protein to ≥ 25% above the lowest response level for 24-hour excretion with an absolute increase of at least 200mg/24 hours of urine M-protein to qualify as "progression"
     * Increase in bone marrow plasma cell percentage to ≥ 25% from lowest response value (the absolute % increase must be ≥ 10%)
  2. Any of the following felt related to the underlying clonal plasma cell proliferative disorder:
     * Hypercalcemia (> 11 mg/dL)
     * Decrease in hemoglobin of ≥ 2 gms/dL
     * Serum creatinine level ≥ 2mg/dL
     * Development of myeloma bone lesions or soft tissue plasmacytoma
Time Frame: Assessed every 3 months for 2 years
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Number analyzed (Participants) | 90 | 92
proportion of participants | 0.93 [0.88 to 0.99] | 0.76 [0.66 to 0.87]
Statistical Analysis 1: Comparison: Arm A (Lenalidomide; Phase III) vs Arm B (Observation; Phase III); Test type: Superiority; p = 0.0005, Log Rank; stratified 1-sided log-rank test

3. Secondary Outcome: Proportion of Participants With Response (Phase II Secondary Endpoint)
Description: Response is defined as complete response (CR), very good partial response (VGPR) or partial response (PR).
  CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-component plus urine M-component < 100 mg per 24 hours
  PR:
  * ≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours
  * If followed by free light chain (FLC) only, a ≥ 50% decrease in the difference between involved and uninvolved FLC levels
  * If unmeasurable disease by serum M-protein, urine M-protein, and serum FLC at baseline, a ≥50% reduction in plasma cells provided baseline bone marrow percentage was ≥ 30%
  * If present at baseline, a ≥ 50% reduction in the size of soft tissue plasmacytomas
Time Frame: Assessed every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, then annually for years 6-10
Population: All registered patients in the phase II part
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase II)
Number analyzed (Participants) | 44
proportion of participants | 0.477 [0.325 to 0.633]

4. Secondary Outcome: Proportion of Participants With Response (Phase III Secondary Endpoint)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Among randomized patients who received treatment or observation
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Number analyzed (Participants) | 88 | 86
proportion of participants | 0.50 [0.391 to 0.608] | 0 [0 to 0.042]

5. Secondary Outcome: 1-year Progression-free Survival (PFS) Rate (Phase III Secondary Endpoint)
Description: PFS is defined as time from randomization to progression or death, whichever occurs first. Patients are considered to have progression if both of the following criteria are met. Kaplan-Meier method was used to estimate 1-year PFS rate.
  1. Any of the following:
     * Increase in serum M-protein to ≥ 25% above the lowest response level with an absolute increase of at least 0.5g/dl to qualify as "progression"
     * Increase in urine M-protein to ≥ 25% above the lowest response level for 24-hour excretion with an absolute increase of at least 200mg/24 hours of urine M-protein to qualify as "progression"
     * Increase in bone marrow plasma cell percentage to ≥ 25% from lowest response value (the absolute % increase must be ≥ 10%)
  2. Any of the following felt related to the underlying clonal plasma cell proliferative disorder:
     * Hypercalcemia (> 11 mg/dL)
     * Decrease in hemoglobin of ≥ 2 gms/dL
     * Serum creatinine level ≥ 2mg/dL
     * Development of myeloma bone lesions or soft tissue plasmacytoma
Time Frame: Assessed every 3 months for one year
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Number analyzed (Participants) | 90 | 92
proportion of participants | 0.98 [0.95 to 1.00] | 0.89 [0.82 to 0.96]

6. Secondary Outcome: 2-year Progression-free Rate (Phase III Secondary Endpoint)
Description: TTP is defined as the time from randomization to progression. Patients are considered to have progression if both of the following criteria are met. Kaplan-Meier method was used to estimate 2-year progression-free rate.
  1. Any of the following:
     * Increase in serum M-protein to ≥ 25% above the lowest response level with an absolute increase of at least 0.5g/dl to qualify as "progression"
     * Increase in urine M-protein to ≥ 25% above the lowest response level for 24-hour excretion with an absolute increase of at least 200mg/24 hours of urine M-protein to qualify as "progression"
     * Increase in bone marrow plasma cell percentage to ≥ 25% from lowest response value (the absolute % increase must be ≥ 10%)
  2. Any one or more of the following felt related to the underlying clonal plasma cell proliferative disorder:
     * Hypercalcemia (> 11 mg/dL)
     * Decrease in hemoglobin of ≥ 2 gms/dL
     * Serum creatinine level ≥ 2mg/dL
     * Development of myeloma bone lesions or soft tissue plasmacytoma
Time Frame: Assessed every 3 months for 2 years
Population: All randomized patients in the phase III part of the study
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Number analyzed (Participants) | 90 | 92
proportion of participants | 94.3 [85.4 to 97.9] | 75.8 [63.6 to 84.4]

7. Secondary Outcome: 2-year Overall Survival (OS) Rate (Phase III Secondary Endpoint)
Description: Overall survival is defined as the time from randomization to death or date last known alive among all randomized patients in the phase III part of the study. Kaplan-Meier method was used to estimate the 2-year OS rate.
Time Frame: Assessed every 3 months for 2 years
Population: All randomized patients in the phase III part of the study
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
Number analyzed (Participants) | 90 | 92
proportion of participants | 0.98 [0.95 to 1.00] | 1.00 [1.00 to 1.00]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 10 years
Description: Serious adverse events are defined as treatment-related adverse events of grade 3 or higher. Other adverse events are treatment-related adverse events not included in serious adverse events.
  Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Arm/Group | Arm A (Lenalidomide; Phase II) | Arm A (Lenalidomide; Phase III) | Arm B (Observation; Phase III)
All-Cause Mortality (participants affected / at risk) | 7/44 | 2/90 | 4/92
Serious Adverse Events (participants affected / at risk) | 23/44 | 40/88 | 8/86
Other Adverse Events (participants affected / at risk) | 14/44 | 20/88 | 5/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Lenalidomide; Phase II) (N=44) | Arm A (Lenalidomide; Phase III) (N=88) | Arm B (Observation; Phase III) (N=86)
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 5 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 7 | 12 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Weight loss (Investigations) | 1 | 1 | 0
White blood cell decreased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2
Thromboembolic event (Vascular disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Lenalidomide; Phase II) (N=44) | Arm A (Lenalidomide; Phase III) (N=88) | Arm B (Observation; Phase III) (N=86)
Anemia (Blood and lymphatic system disorders) | 6 | 5 | 2
Fatigue (General disorders) | 4 | 9 | 2
Constipation (Gastrointestinal disorders) | 2 | 7 | 1
Lymphocyte count decreased (Investigations) | 3 | 4 | 2
Neutrophil count decreased (Investigations) | 5 | 8 | 1
Platelet count decreased (Investigations) | 5 | 5 | 1
White blood cell decreased (Investigations) | 6 | 9 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT01169337/Prot_SAP_000.pdf